CLINICAL TRIAL: NCT05081765
Title: The Effect of Glucose Level and Diabetes Mellitus on the Plasma Minimum Steady-state Concentration Ctrough of Olaparib in Patients With Ovarian Cancer
Brief Title: The Effect of Glucose Level and Diabetes Mellitus on Ctrough of Olaparib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Poznan University Hospital of Lord's Transfiguration (Other)
Responsible Party: Principal Investigator, Stanisławiak-Rudowicz Joanna, Principal Investigator, Clinical Doctor, Poznan University of Medical Sciences
Other Study IDs: 697/20
Record Dates: First submitted 2021-10-01; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Ovary Cancer
Keywords: olaparib; blood-level testing; C through; diabetes melitus; hyperglycemia
MeSH Terms: conditions — Ovarian Neoplasms; Hyperglycemia | interventions — olaparib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — The probe with blood taken to check the C through of olaparib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Patients with diabetes mellitus: olaparib 2 x 300mg /24h tablets = olaparib 2 x 400mg/24 olaparib 2 x 250mg/24h tablets = olaparib 2 x 200mg/24h olaparib 2 x 200mg/24h tablets = olaparib 2 x 100mg/24h
  Interventions: Drug: Lynparza® (AstraZeneca Pharma Poland Sp. z o.o.); Device: Lynparza
- Patients with hyperglycemia,: olaparib 2 x 300mg /24h tablets = olaparib 2 x 400mg/24 olaparib 2 x 250mg/24h tablets = olaparib 2 x 200mg/24h olaparib 2 x 200mg/24h tablets = olaparib 2 x 100mg/24h
  Interventions: Drug: Lynparza® (AstraZeneca Pharma Poland Sp. z o.o.); Device: Lynparza
- Patient with normal glucose level: olaparib 2 x 300mg /24h tablets = olaparib 2 x 400mg/24 olaparib 2 x 250mg/24h tablets = olaparib 2 x 200mg/24h olaparib 2 x 200mg/24h tablets = olaparib 2 x 100mg/24h
  Interventions: Drug: Lynparza® (AstraZeneca Pharma Poland Sp. z o.o.); Device: Lynparza

INTERVENTIONS:
Drug: Lynparza® (AstraZeneca Pharma Poland Sp. z o.o.) — correlation between C through and taken drug
  Other Names: olaparib
Device: Lynparza — correlation between C through and taken drug
  Other Names: olaparib

SUMMARY:
Monitored therapy of olaparib concentrations in the blood of diabetic population probably will assess the need for individual dosing of the drug.

The project concerns on the monitored therapy of olaparib in a population of patients with DM, hyperglycemia and normal glucose level.

Currently, there are no studies assessing the effect of comorbidities and of the administered drugs on the pharmacokinetics of olaparib.

DETAILED DESCRIPTION:
The research is conducted at the Poznan University of Medical Sciences, and the Poznan, Poland with the approval from the Bioethics Committee, University of Medical Sciences, Poznan, Poland (697/20). The subjects of the research: the C through of olaparib in the patients with ovarian cancer who received olaparib The patients included in the study if they met the following criteria: treatment with olaparib above four days, age >18 years; no history of allergy to olaparib. The chief criteria for exclusion included allergy to olaparib, age under 18 years, status of the patient which do not allowed the patient to continue the study.

Administration and blood sampling The patients with an ovarian cancer treated with olaparib (tablets in dose 300mg/12h, 250mg/12h, 200 mg/12h or capsules 400mg/12h, 200mg/12h, 100 mg/12h).

Blood samples (2 mL) collected at steady state before morning drug administration. The blood samples transferred into heparinised tubes and centrifuged at 2880 g for 10 min at 4 °C. Next the plasma transferred to propylene tubes and stored at - 20 °C until analysis.

Assays The concentrations of olaparib in plasma assayed using the high-performance liquid chromatography (HPLC) method with ultraviolet (UV) detection. The method validated according to European Medicines Agency guideline. The method validation confirmed good precision (CV% <15%), accuracy (92.3-115.0%) and linearity (r=0.9994) in the range of 100-4000 ng/mL.

The severity of olaparib adverse effects assessed by CTCAE (Common Terminology Criteria for Adverse Events) v.5.0 scale.

ELIGIBILITY:
Inclusion Criteria:

* ovarian cancer patients treated with olaparib above than 4 days
* patient who gave permission to take part in the trial
* age >18 years
* no history of allergy to olaparib

Exclusion Criteria:

* allergy to olaparib,
* age under 18 years,
* status of the patient which do not allowed the patient to continue the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of the research are patients with ovarian cancer who received olaparib as a maintance therapy after platin basen chemotherapy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation between glucose level and C through.olaparib in the blood of the patients with ovarian cancer | through study completion, an average of 1 year
  There is idea to check the correlation of C through of the olaparib taken by the patients with diabetes melitus and ovarian cancer and the correlation of C through and glucose of the patients with hyperglycemia diagnosed during olaparib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joanna J Stanisławiak - Rudowicz, Principal Investigator — University of Medical Sciences Poznań, Poland
Locations (1):
- University od Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
To check C through of olaparib and morphology, Alat, Aspat and GFR and glucose level

REFERENCES:
- [Background] Debska S, Kubicka J, Czyzykowski R, Habib M, Potemski P. [PARP inhibitors--theoretical basis and clinical application]. Postepy Hig Med Dosw (Online). 2012 May 30;66:311-21. doi: 10.5604/17322693.999033. Polish. PMID 22706117
- [Background] Wisnik E, Ryksa M, Koter-Michalak M. [PARP1 inhibitors: contemporary attempts at their use in anticancer therapy and future perspective]. Postepy Hig Med Dosw (Online). 2016 Apr 13;70:280-94. doi: 10.5604/17322693.1199303. Polish. PMID 27117104
- [Background] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott CL, Meier W, Shapira-Frommer R, Safra T, Matei D, Fielding A, Spencer S, Dougherty B, Orr M, Hodgson D, Barrett JC, Matulonis U. Olaparib maintenance therapy in patients with platinum-sensitive relapsed serous ovarian cancer: a preplanned retrospective analysis of outcomes by BRCA status in a randomised phase 2 trial. Lancet Oncol. 2014 Jul;15(8):852-61. doi: 10.1016/S1470-2045(14)70228-1. Epub 2014 May 31. PMID 24882434
- [Background] Friedlander M, Banerjee S, Mileshkin L, Scott C, Shannon C, Goh J. Practical guidance on the use of olaparib capsules as maintenance therapy for women with BRCA mutations and platinum-sensitive recurrent ovarian cancer. Asia Pac J Clin Oncol. 2016 Dec;12(4):323-331. doi: 10.1111/ajco.12636. PMID 27917619
- [Background] Szalek E, Karbownik A, Sobanska K, Grabowski T, Polom W, Lewandowska M, Wolc A, Matuszewski M, Grzeskowiak E. The pharmacokinetics and hypoglycaemic effect of sunitinib in the diabetic rabbits. Pharmacol Rep. 2014 Oct;66(5):892-6. doi: 10.1016/j.pharep.2014.05.011. Epub 2014 Jun 6. PMID 25149997
- [Background] Karbownik A, Szalek E, Sobanska K, Grabowski T, Wolc A, Grzeskowiak E. The alteration of pharmacokinetics of erlotinib and OSI420 in type 1 diabetic rabbits. Pharmacol Rep. 2016 Oct;68(5):964-8. doi: 10.1016/j.pharep.2016.04.015. Epub 2016 May 6. PMID 27372922
- [Background] Dostalek M, Court MH, Yan B, Akhlaghi F. Significantly reduced cytochrome P450 3A4 expression and activity in liver from humans with diabetes mellitus. Br J Pharmacol. 2011 Jul;163(5):937-47. doi: 10.1111/j.1476-5381.2011.01270.x. PMID 21323901
- [Background] Dostalek M, Akhlaghi F, Puzanovova M. Effect of diabetes mellitus on pharmacokinetic and pharmacodynamic properties of drugs. Clin Pharmacokinet. 2012 Aug 1;51(8):481-99. doi: 10.2165/11631900-000000000-00000. PMID 22668340
- [Background] Tran M, Elbarbry F. Influence of diabetes mellitus on pharmacokinetics of drugs. MOJ Bioequiv Availab. 2016;2(1):3-4.
- [Background] Porazka J, Szalek E, Polom W, Czajkowski M, Grabowski T, Matuszewski M, Grzeskowiak E. Influence of Obesity and Type 2 Diabetes Mellitus on the Pharmacokinetics of Tramadol After Single Oral Dose Administration. Eur J Drug Metab Pharmacokinet. 2019 Aug;44(4):579-584. doi: 10.1007/s13318-019-00543-1. PMID 30778911
- [Background] Stachowiak A, Szalek E, Karbownik A, Lojko A, Porazka J, Przewozna I, Grabowski T, Wolc A, Grzeskowiak E. The Influence of Diabetes Mellitus on Glucuronidation and Sulphation of Paracetamol in Patients with Febrile Neutropenia. Eur J Drug Metab Pharmacokinet. 2019 Apr;44(2):289-294. doi: 10.1007/s13318-018-0508-4. PMID 30187443
- [Background] Karbownik A, Szalek E, Sobanska K, Klupczynska A, Plewa S, Grabowski T, Wolc A, Moch M, Kokot ZJ, Grzeskowiak E. A pharmacokinetic study on lapatinib in type 2 diabetic rats. Pharmacol Rep. 2018 Apr;70(2):191-195. doi: 10.1016/j.pharep.2017.09.003. Epub 2017 Sep 18. PMID 29471066
- [Background] Karbownik A, Stachowiak A, Urjasz H, Sobanska K, Szczecinska A, Grabowski T, Stanislawiak-Rudowicz J, Wolc A, Grzeskowiak E, Szalek E. The oxidation and hypoglycaemic effect of sorafenib in streptozotocin-induced diabetic rats. Pharmacol Rep. 2020 Feb;72(1):254-259. doi: 10.1007/s43440-019-00021-0. Epub 2020 Jan 8. PMID 32016844
- See also: Summary of product characteristic — https://www.ema.europa.eu/en/documents/product-information/lynparza-epar-product-information_pl.pdf
- See also: Onkol Prakt Klin Edu 2018;4(3):167-178. — https://journals.viamedica.pl/onkologia_w_praktyce_klin_edu/article/view/58916